CLINICAL TRIAL: NCT06677463
Title: An Evaluation of Virtual Reality in Labor Pain During Vaginal Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Amgad Hamed Abo motaa, physical therapy specialist for women health, Kafrelsheikh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KFS IRB200-91
Record Dates: First submitted 2024-10-30; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: An Evaluation of Virtual Reality in Labor Pain During Vaginal Childbirth

STUDY DESIGN:
Intervention Model Description: This study will be conducted to evaluate the effect of applying virtual reality among laboring women during first stage of labor
Masking Description: This study will be conducted to evaluate the effect of applying virtual reality among laboring women during first stage of labor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- An experimental study on the effect of virtual reality glasses on women during childbirth (Experimental): An experimental study on the effect of virtual reality glasses on women during childbirth
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Studying the effect of virtual reality glasses on women during pregnancy, for the first time, it is also used to facilitate the birth process

SUMMARY:
This study will be conducted to evaluate the effect of applying virtual reality among laboring women during first stage of labor

DETAILED DESCRIPTION:
This study will be conducted to evaluate the effect of applying virtual reality among laboring women during first stage of labor

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-25 years old .
* body mass index (BMI) 25- 32 kg/m2 .
* Primiparous .
* Highly educated.

Exclusion Criteria:

* Laboring women with high risk pregnancy.
* Laboring women are taking pharmacological methods to relieve pain during first stage of labor.
* Low educated women

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The pregnant woman during normal labor
Enrollment: 80 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Serum cortisol levels | Immediately after the intervention
  Serum cortisol levels during the normal labor
Time of labor | Immediately after the intervention
  Measure the time of labor after delivery
Type of labor normal , cesarean section or episiotomy | Immediately after the intervention
  Type of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Fayiz Elshamy Elshamy Fayiz Elshamy, Professor of physical therapy, Principal Investigator — Fayiz Elshamy
Locations (1):
- Menshawy general hospital, Tanta, Gharabia, Egypt

IPD SHARING:
Plan to Share IPD: No
These pregnant women were asked to bring their phone that the video was recorded with them to the labour. When the pregnant women got into labour, they would hospitalized . The follow-ups and labour will also performed . These two-dimensional images will converted into three-dimensional images through an application installed in the mother's phone and will showe to her with a VR Box 3D virtual reality glass one after another. In cases where the program was not compatible with the mother's phone, it will watched on the researcher's phone. The total duration of image viewing was recorded. Procedure of application of virtual reality from cervical dilatation 3 cm to full dilatation